CLINICAL TRIAL: NCT04532619
Title: A Pilot Study of the Fathering Through Change Intervention for Fathers With Substance Use Disorders
Brief Title: A Substance Use Adaptation of Fathering Through Change
Acronym: FTC-SUD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oregon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 12132019.029
Record Dates: First submitted 2020-07-22; First posted 2020-08-31 (Actual); Results first posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2022-03

CONDITIONS: Parenting; Substance Use
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): 6 weeks of Fathering Through Change videos and 3 individual coaching calls.
  Interventions: Behavioral: Fathering Through Change
- Control (No Intervention): Links to parenting websites

INTERVENTIONS:
Behavioral: Fathering Through Change — Fathering Through Change is an adaptation of Parent Management Training Oregon. This pilot provides a limited version of Fathering Through Change via text messaged and emailed weekly video content and includes individual coaching calls.
  Arms: Intervention

SUMMARY:
This study is a randomized control trial of the Fathering Through Change intervention, delivered via text messaging, to fathers in recovery for substance use disorders.

ELIGIBILITY:
Inclusion Criteria:

* identify as being in recovery
* abstinent from illicit substances for at least 1 day and less than one year at time of enrollment
* parenting responsibilities for a child between the ages of 3-16
* spend at least 2 hours per week with child between ages of 3-16
* English speaking

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Must identify as a father.
Enrollment: 41 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Camille C Cioffi, PhD, Study Director — University of Oregon
Locations (1):
- Willamette Family Treatment Center, Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared with the Center on Parenting and Opioids in a repository. The data repository will initially be available only to Center on Parenting and Opioids investigators and will later become accessible for other researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The Center on Parenting and Opioids will determine the data's availability.
Access Criteria: Initially only to Center on Parenting and Opioids researchers. Future public access will be determined by the Center on Parenting and Opioids (PI: Leve)

REFERENCES:
- [Background] DeGarmo DS, Jones JA. Fathering Through Change (FTC) intervention for single fathers: Preventing coercive parenting and child problem behaviors. Dev Psychopathol. 2019 Dec;31(5):1801-1811. doi: 10.1017/S0954579419001019. PMID 31489831
- [Derived] Cioffi CC, Browning O'Hagan AM, Halvorson S, DeGarmo DS. A randomized controlled trial to improve fathering among fathers with substance use disorders: Fathering in recovery intervention. J Fam Psychol. 2023 Dec;37(8):1303-1314. doi: 10.1037/fam0001134. Epub 2023 Sep 11. PMID 37695329

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited from substance use disorder treatment centers
Pre-assignment Details: No pre-assignment details to report
Period: Overall Study
Arm/Group | Intervention | Control
Started | 21 | 20
Completed | 18 | 19
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 21 | 20 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 20 | 41
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 40 [35 to 45] | 35 [33 to 42] | 39 [34 to 45]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 21 | 20 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 7
  Not Hispanic or Latino | 18 | 16 | 34
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 0 | 3 | 3
  White | 17 | 11 | 28
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 2 | 3 | 5
TOPSE: Parenting Self-Efficacy [Median (Inter-Quartile Range); unit: units on a scale] — The Tool to Measure Parenting Self-Efficacy (TOPSE) consists of 48 self-efficacy statements. There are six self-efficacy statements for each domain and parents indicate how much they agree with each statement by responding to a Likert scale from 0-10 where 0 equates to completely disagree and 10 equates to completely agree. We administered the play, acceptance, and control domains. The overall score (0-10) was computed as the mean of these three sub-scale means. A higher overall score indicates greater self-efficacy.
  units on a scale | 7.78 [7.53 to 9.01] | 7.87 [7.24 to 8.44] | 7.78 [7.28 to 8.58]
Parenting Practices: Harsh parenting [Median (Inter-Quartile Range); unit: units on a scale] — The Parenting Practices Interview is a standardized instrument to measure parenting skills. The harsh parenting sub-scale is computed as the average (1-7) of 6 items. Lower scores are more desirable. Population: Complete scores
  units on a scale
    number analyzed (Participants) | 20 | 20 | 40
    (all) | 2.08 [1.5 to 3] | 2.17 [1.63 to 2.67] | 2.17 [1.5 to 2.88]
Parenting Practices: Inept parenting [Median (Inter-Quartile Range); unit: units on a scale] — Parenting Practices Interview is a standardized instrument to measure parenting skills. The inept parenting sub-scale is computed as the average (1-7) of 11 items. Lower scores are more desirable. Population: Complete scores
  units on a scale
    number analyzed (Participants) | 20 | 20 | 40
    (all) | 2.5 [2.23 to 2.86] | 3.00 [2.43 to 3.39] | 2.64 [2.27 to 3.11]
Parenting Practices: Prosocial parenting [Median (Inter-Quartile Range); unit: units on a scale] — Parenting Practices Interview is a standardized instrument to measure parenting skills. The prosocial parenting sub-scale is computed as the average (1-7) of 15 items. Higher scores are more desirable. Population: Complete scores
  units on a scale
    number analyzed (Participants) | 20 | 20 | 40
    (all) | 4.87 [4.13 to 5.2] | 4.27 [4.03 to 4.68] | 4.60 [4.07 to 5.07]
Substance Use: Any Use in the Last 30 Days [Count of Participants; unit: Participants] — Substance use is collected using the Center on Parenting and Opioids substance use questionnaire. We measured substance use as a dichotomous variable: any use of alcohol, cannabis, and illicit substances in the past thirty days. Population: Non-missing values
  Participants
    number analyzed (Participants) | 20 | 20 | 40
    (all) | 4 | 7 | 11
Substance Use: Days of Use the Last 30 [Median (Inter-Quartile Range); unit: Days] — Substance use is collected using the Center on Parenting and Opioids substance use questionnaire. We measured substance use continuous variable: number of days using of alcohol, cannabis, and illicit substances in the past thirty days.
  Days | 0 [0 to 0] | 0 [0 to 16] | 0 [0 to 2]
Child Behavior: Strengths and Difficulties Questionnaire [Median (Inter-Quartile Range); unit: units on a scale] — Child behavior as measured by the Strengths and Difficulties Questionnaire overall score. This scale includes twenty-five items rated on a 3-point scale ranging from 0 to 2. There are five sub-scales each composed of 5 items: emotional regulation, conduct, hyperactivity, peer problems, and prosocial behavior. The prosocial sub-scale was not used for analyses and the twenty items remaining were summed into an overall score (0-40). Higher scores are more desirable. Population: Complete scores
  units on a scale
    number analyzed (Participants) | 20 | 20 | 40
    (all) | 11 [8 to 17] | 11 [7 to 14] | 11 [8 to 15]

OUTCOME MEASURES:

1. Primary Outcome: TOPSE: Group Mean Change at 6 Weeks and 4 Months on the Tool of Parenting Self-Efficacy
Description: The Tool to Measure Parenting Self-Efficacy (TOPSE) consists of 48 self-efficacy statements. There are six self-efficacy statements for each domain and parents indicate how much they agree with each statement by responding to a Likert scale from 0-10 where 0 equates to completely disagree and 10 equates to completely agree. We administered the play, acceptance, and control domains. The overall score (0-10) was computed as the mean of these three sub-scale means. A higher overall score indicates greater self-efficacy.
Time Frame: baseline to 6 weeks and baseline to 4 months
Population: Overall number analyzed is the number of participants with at least one follow-up.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 18 | 19
score on a scale
  6 weeks: number analyzed (Participants) | 17 | 18
  6 weeks | 8.77 [7.84 to 9.32] | 7.50 [7.10 to 8.53]
  4 months: number analyzed (Participants) | 17 | 17
  4 months | 8.70 [7.96 to 9.38] | 7.65 [7.22 to 8.33]
Statistical Analysis 1: Comparison: Intervention vs Control; We used a multilevel models to produce regression estimates. We used multiple imputation. Intervention enrollment was coded as 1 and enrollment in the control arm was coded as 0. We accounted for baseline values and psychopathology; Test type: Superiority; p = 0.014, Mixed Models Analysis — Computed p-value; Slope = .5, 95% CI 2-sided [0.10 to 0.89]

2. Primary Outcome: PPI Harsh: Group Mean Change at 6 Weeks and 4 Months the Parenting Practices Interview Harsh Parenting Subscale
Description: The Parenting Practices Interview is a standardized instrument to measure parenting skills. The harsh parenting sub-scale is computed as the average (1-7) of 6 items. Lower scores are more desirable.
Time Frame: baseline to 6 weeks and baseline to 4 months
Population: Overall number analyzed is the number of participants with at least one follow-up.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 18 | 19
units on a scale
  6 weeks: number analyzed (Participants) | 17 | 18
  6 weeks | 1.67 [1.33 to 2.83] | 2.08 [1.71 to 2.62]
  4 months: number analyzed (Participants) | 17 | 17
  4 months | 1.83 [1.33 to 2.00] | 2.00 [1.50 to 2.83]
Statistical Analysis 1: Comparison: Intervention vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.80, Mixed Models Analysis — computed p-value; Slope = -0.05, 95% CI 2-sided [-0.41 to 0.32]

3. Primary Outcome: PPI Inept: Group Mean Change at 6 Weeks and 4 Months the Parenting Practices Interview Inept Parenting Subscale
Description: Parenting Practices Interview is a standardized instrument to measure parenting skills. The inept parenting sub-scale is computed as the average (1-7) of 11 items. Lower scores are more desirable.
Time Frame: baseline to 6 weeks and baseline to 4 months
Population: Overall number analyzed is the number of participants with at least one follow-up.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 18 | 19
units on a scale
  6 weeks: number analyzed (Participants) | 17 | 18
  6 weeks | 2.09 [1.91 to 2.82] | 2.91 [2.68 to 3.55]
  4 months: number analyzed (Participants) | 17 | 17
  4 months | 2.09 [1.73 to 2.64] | 2.64 [2.27 to 3.18]
Statistical Analysis 1: Comparison: Intervention vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.009, Mixed Models Analysis — computed p-value; Slope = -0.29, 95% CI 2-sided [-0.51 to -0.07]

4. Primary Outcome: PPI Prosocial: Group Mean Change at 6 Weeks and 4 Months the Parenting Practices Interview Prosocial Parenting Subscale
Description: Parenting Practices Interview is a standardized instrument to measure parenting skills. The prosocial parenting subscale is computed as the mean of 15 items on all rated on a 1-7 scale. Higher scores are more desirable.
Time Frame: baseline to 6 weeks and baseline to 4 months
Population: Overall number analyzed is the number of participants with at least one follow-up.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 18 | 19
units on a scale
  6 weeks: number analyzed (Participants) | 17 | 18
  6 weeks | 5.07 [4.67 to 5.40] | 4.33 [4.17 to 4.77]
  4 months: number analyzed (Participants) | 17 | 17
  4 months | 4.93 [4.60 to 5.40] | 4.80 [4.07 to 5.00]
Statistical Analysis 1: Comparison: Intervention vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.118, Mixed Models Analysis — calculated p-value; Slope = 0.17, 95% CI 2-sided [-0.04 to 0.38]

5. Secondary Outcome: Substance Use: Group Mean Change at 6 Weeks and 4 Months on Any Use in the Last 30 Days
Description: Substance use is collected using the Center on Parenting and Opioids substance use questionnaire. We measured substance use as a dichotomous variable: any use of alcohol, cannabis, and illicit substances in the past thirty days.
Time Frame: baseline to 6 weeks and baseline to 4 months
Population: Number analyzed is the number of participants with at least one follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 18 | 19
Participants
  6 weeks: number analyzed (Participants) | 17 | 18
  6 weeks | 4 | 6
  4 months: number analyzed (Participants) | 17 | 17
  4 months | 4 | 8
Statistical Analysis 1: Comparison: Intervention vs Control; We used a multilevel models to produce regression estimates. We used multiple imputation. Intervention enrollment was coded as 1 and enrollment in the control arm was coded as 0. We accounted for baseline values and psychopathology. A logistic link function was used for this binary outcome; Test type: Superiority; p = .24, Mixed Models Analysis — computed p-value; Odds Ratio, log = -0.90, Standard Error of Mean .77

6. Secondary Outcome: Substance Use: Group Mean Change at 6 Weeks and 4 Months on Days of Use the Last 30
Description: Substance use is collected using the Center on Parenting and Opioids substance use questionnaire. We measured substance use count variable: number of days using of alcohol, cannabis, and illicit substances in the past thirty days.
Time Frame: baseline to 6 weeks and baseline to 4 months
Population: Number analyzed is the number of participants with at least one follow-up.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Intervention | Control
Number analyzed (Participants) | 18 | 19
days
  6 weeks | 0 [0 to 0] | 0 [0 to 2.50]
  4 months | 0 [0 to 0] | 0 [0 to 15]
Statistical Analysis 1: Comparison: Intervention vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.43, Mixed Models Analysis — computed p-value; Slope = -1.33, 95% CI 2-sided [-4.64 to 1.98]

7. Secondary Outcome: SDQ: Group Mean Change at 4 Months on Child Behavior
Description: Child behavior as measured by the Strengths and Difficulties Questionnaire overall score. This scale includes twenty-five items rated on a 3-point scale ranging from 0 to 2. There are five subscales each composed of 5 items: emotional regulation, conduct, hyperactivity, peer problems, and prosocial behavior. The prosocial scale was not used for analyses and the twenty items remaining were summed into an overall score (0-40). Higher scores are more desirable.
Time Frame: baseline to 4 months
Population: Overall number analyzed is the number of participants with at least one follow-up.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 16 | 16
units on a scale | 9 [4.5 to 11] | 16 [6.75 to 21]
Statistical Analysis 1: Comparison: Intervention vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.07, Mixed Models Analysis — computed p-value; Slope = -2.06, 95% CI 2-sided [-4.27 to 0.15]

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/20
Other Adverse Events (participants affected / at risk) | 0/21 | 0/20

LIMITATIONS AND CAVEATS:
This was an underpowered randomized controlled trial. The purpose of the study was to assess feasibility of the Fathering In Recovery intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (3):
  • Study Protocol (2021-07-08): https://cdn.clinicaltrials.gov/large-docs/19/NCT04532619/Prot_001.pdf
  • Statistical Analysis Plan (2023-03-19): https://cdn.clinicaltrials.gov/large-docs/19/NCT04532619/SAP_002.pdf
  • Informed Consent Form (2020-10-15): https://cdn.clinicaltrials.gov/large-docs/19/NCT04532619/ICF_003.pdf